CLINICAL TRIAL: NCT00808600
Title: Empowerment of Lung and Heart-lung Transplant Patients by a Multimodal Resource-activating Behavioural Training Programme and Cardiopulmonary Exercise - a Randomised Controlled Study
Brief Title: Empowerment of Lung and Heart-lung Transplant Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Prof. Dr. Harald Guendel, Department of Psychosomatics and Psychotherapy, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFB-application 32
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Lung Transplantation; Heart-Lung Transplantation; "Rehabilitation"; Psychotherapy; Exercise Training
Keywords: lung transplantation; heart-lung transplantation; rehabilitation; resource-activating training; anaerobic exercise training
MeSH Terms: interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- resource-activating training, intensified exercise training (Other): combination of the two interventions: resource-activating behavioural training and intensified exercise training
  Interventions: Behavioral: resource-activating behavioural training programme; Behavioral: Intensified anaerobic exercise training
- resource-activating training, moderate exercise training (Other): combination of the two interventions: resource-activating training and moderate exercise training
  Interventions: Behavioral: resource-activating behavioural training programme; Behavioral: Moderate aerobic exercise training
- relaxation training, intensified exercise training (Other): combination of the two interventions: relaxation training and intensified exercise training
  Interventions: Behavioral: Relaxation training; Behavioral: Intensified anaerobic exercise training
- relaxation training, moderate exercise training (Other): combination of the two interventions: relaxation training and moderate exercise training
  Interventions: Behavioral: Relaxation training; Behavioral: Moderate aerobic exercise training

INTERVENTIONS:
Behavioral: resource-activating behavioural training programme — Stepwise intervention based on the principles of resource-activating training (RAT) applied to the needs of patients in the process after lung transplantation.
  Phase 1: Build-up of therapeutic relationship through resource-activating training for patients after transplantation during rehabilitation in the rehabilitation centre Fallingbostel following inpatient treatment. Phase 2: Continued resource-activation and transfer by means of internet-based interventions (1 per 2 weeks) as well as personal interventions by trained nurses and a clinical psychologist during regular out-patient visits (approx. 4 times per year) over one year immediately following rehabilitation. Interventions focus on strengthening individual and interpersonal resources for well-being, psychoeducation, stress management and coping with illness. Phase 3: Termination and transfer, including a detailed medical report.
  Arms: resource-activating training, intensified exercise training; resource-activating training, moderate exercise training
Behavioral: Relaxation training — Phase 1: Build-up of therapeutic relationship through resource-activating training for patients after transplantation during rehabilitation in the rehabilitation centre Fallingbostel following inpatient treatment. Phase 2: Regular relaxation training after rehabilitation by self-guided relaxation compact disk and accompanying worksheets.
  Arms: relaxation training, intensified exercise training; relaxation training, moderate exercise training
Behavioral: Intensified anaerobic exercise training — Phase 1: Recruitment and initiation of intensified and individualised aerobic/anaerobic exercise training based on determination of aerobic/anaerobic threshold during rehabilitation in the rehabilitation centre Fallingbostel. During rehabilitation daily training sessions with a duration of 30 minutes each are performed under medical supervision. Phase 2: Home training on an IT-assisted ergometer 3.5 times a week with interval exercise intensity above the anaerobic threshold. Work load and heart rate are stored by an ergometer-chip, lung function analyses are performed and should be transferred via phone-based telemetry. Exercise training intensities will be adapted monthly, corresponding to training results. At regular 3 months visits to the outpatient clinic a medical examination is carried out. Moreover, according to the actual functional state of the patient estimated 3 monthly training work load will be adjusted. Phase 3: Termination, evaluation after a period of 12 months.
  Arms: relaxation training, intensified exercise training; resource-activating training, intensified exercise training
Behavioral: Moderate aerobic exercise training — Phase 1: Recruitment and initiation of moderate aerobic exercise training based on 40 percent of maximal oxygen consumption in Watt during rehabilitation in the rehabilitation centre Fallingbostel. Phase 2: Moderate aerobic endurance training with the target intensity of 40 percent of the individual maximum exercise capacity will be performed 3.5 times a week with a duration of 30 minutes per session, work load will be adapted continuously according to the measures that are assessed during the repeated control examinations after periods of 3 months in the outpatient clinic of the pulmonary department of Hanover Medical School.
  Arms: relaxation training, moderate exercise training; resource-activating training, moderate exercise training

SUMMARY:
Lung or combined heart-lung transplantation represents an established treatment strategy for patients with end-stage lung disease. Transplantation results in an increased exercise capacity, a better quality of life and - depending on the pulmonary disease - a prolonged life compared to the natural course of the pulmonary disease. However, even after successful organ transplantation, patients realise the often inflated, unrealistic character of their previous expectations due to their continuing dependence on medication, regular control examinations and a higher risk of infections and allograft rejections. Patients have to cope with erupting demands in family, social and work life. It becomes evident that their lives have changed forever. In this context, limitations in mental health like depression and reduced quality of life (QoL) as well as diminished compliance may emerge or even persist. By five years post-transplant, about one-half of the patients meet the criteria of an anxiety disorder. Symptoms of a clinically relevant depression or mood disorder occur in 10 to 15 % of lung transplant patients.

In addition, patients after lung transplantation are often in a poor physical condition and only hold a reduced functional status. Surgery itself, a prolonged weaning period during mechanical ventilation, sepsis, and especially the immunosuppressive medication may long-ranging or permanently limit physical activity, further reducing muscle mass and bodily function.

Some positive effects of either psychological coping skills training or supervised exercise therapy after lung or heart-lung transplantation on QoL and functional status have been described in very few existing pilot studies with small numbers of patients and only short-term follow-up. In addition, although clear evidence points to a mutual amplifying effect of both psychological training and exercise therapy in patients coping with chronic disease, no such study has yet been conducted in the transplantation field.

Therefore, the aim of the investigators randomised controlled study is to prove the differential benefit of a multi-modal resource-activating behavioural training programme combined with an intensified exercise training programme on functional status as well as on QoL in a four-armed design. The investigators hypotheses are: (H1) The multimodal resource-activating behavioural training programme will show better out-comes in the measures of global health-related QoL compared to a relaxation group. (H2) Participants in the intensified anaerobic exercise training will have better outcomes in the measures of exercise-related variables and lung function than the group with moderate aerobic exercise training. (H3) Participants in the behavioural intervention programme and the intensified exercise training will have better outcomes in the measures of global health-related QoL and exercise-related variables compared to the other groups.

ELIGIBILITY:
Inclusion Criteria:

* All individuals following lung or combined heart-lung transplantation at Hanover Medical School

Exclusion Criteria:

* Severe bronchus stenosis after surgery
* Uncontrolled hypertension
* Orthopedic impairment
* Oxygen desaturation during exercise to less than 89 % without supplemental oxygen
* Cardiovascular complications that limit exercise tolerance
* Persistent multi-drug resistant infections (MRSA, VRE, Burkholderia Cepacia, Pandorea)
* Severe psychiatric disorders

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2009-10; Primary Completion 2013-07 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
SF-36 Physical and Psychological Component Summary | T0: before rehab, T1: after rehab, T2: after intervention phase, T3: after 1-year follow-up
Maximum exercise capacity in Watts absolutely and in percentage predicted and anaerobic threshold | T0: before rehab, T1: after rehab, T2: after intervention phase, T3: after 1-year follow-up
Oxygen uptake per minute and kg body mass [VO2/min/kg/Body weight] absolutely and in percentage predicted | T0: before rehab, T1: after rehab, T2: after intervention phase, T3: after 1-year follow-up
Duration of exercise in minutes during constant load tests in the range of the anaerobic threshold | T0: before rehab, T1: after rehab, T2: after intervention phase, T3: after 1-year follow-up

SECONDARY OUTCOMES:
St. George Respiratory Questionnaire (SGRQ) | T0: before rehab, T1: after rehab, T2: after intervention phase, T3: after 1-year follow-up
Hospital Anxiety and Depression Scale (HADS) | T0: before rehab, T1: after rehab, T2: after intervention phase, T3: after 1-year follow-up
Social Support Questionnaire (F-SozU) | T0: before rehab, T1: after rehab, T2: after intervention phase, T3: after 1-year follow-up
Life Orientation Test (LOT) | T0: before rehab, T1: after rehab, T2: after intervention phase, T3: after 1-year follow-up
Compliance to medical treatment, exercise training, and lung function measurements at patients' home by an asthma monitor | T0: before rehab, T1: after rehab, T2: after intervention phase, T3: after 1-year follow-up
other variables of functional status | T0: before rehab, T1: after rehab, T2: after intervention phase, T3: after 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Harald Gündel, Prof. Dr., Principal Investigator — Dept. of Psychosomatics and Psychotherapy, Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Background] Ambrosino N, Strambi S. New strategies to improve exercise tolerance in chronic obstructive pulmonary disease. Eur Respir J. 2004 Aug;24(2):313-22. doi: 10.1183/09031936.04.00002904. PMID 15332404
- [Background] Blumenthal JA, Babyak MA, Keefe FJ, Davis RD, Lacaille RA, Carney RM, Freedland KE, Trulock E, Palmer SM. Telephone-based coping skills training for patients awaiting lung transplantation. J Consult Clin Psychol. 2006 Jun;74(3):535-44. doi: 10.1037/0022-006X.74.3.535. PMID 16822110
- [Background] De Vito Dabbs A, Hoffman LA, Swigart V, Happ MB, Dauber JH, McCurry KR, Iacono A. Striving for normalcy: symptoms and the threat of rejection after lung transplantation. Soc Sci Med. 2004 Oct;59(7):1473-84. doi: 10.1016/j.socscimed.2004.01.013. PMID 15246175
- [Background] Dew MA, DiMartini AF. Psychological disorders and distress after adult cardiothoracic transplantation. J Cardiovasc Nurs. 2005 Sep-Oct;20(5 Suppl):S51-66. doi: 10.1097/00005082-200509001-00007. PMID 16160585
- [Background] Dew MA, Goycoolea JM, Harris RC, Lee A, Zomak R, Dunbar-Jacob J, Rotondi A, Griffith BP, Kormos RL. An internet-based intervention to improve psychosocial outcomes in heart transplant recipients and family caregivers: development and evaluation. J Heart Lung Transplant. 2004 Jun;23(6):745-58. doi: 10.1016/j.healun.2003.07.002. PMID 15366436
- [Background] Dew MA, Kormos RL, DiMartini AF, Switzer GE, Schulberg HC, Roth LH, Griffith BP. Prevalence and risk of depression and anxiety-related disorders during the first three years after heart transplantation. Psychosomatics. 2001 Jul-Aug;42(4):300-13. doi: 10.1176/appi.psy.42.4.300. PMID 11496019
- [Background] Gimenez M, Servera E, Vergara P, Bach JR, Polu JM. Endurance training in patients with chronic obstructive pulmonary disease: a comparison of high versus moderate intensity. Arch Phys Med Rehabil. 2000 Jan;81(1):102-9. doi: 10.1016/s0003-9993(00)90229-6. PMID 10638884
- [Background] Hentschel M, Becker J, Lepthin HJ. [Effects of a high intensity training program on patients with chronic obstructive airways disease (COAD)]. Pneumologie. 2002 Apr;56(4):240-6. doi: 10.1055/s-2002-25073. German. PMID 11951158
- [Background] Kugler C, Fischer S, Gottlieb J, Welte T, Simon A, Haverich A, Strueber M. Health-related quality of life in two hundred-eighty lung transplant recipients. J Heart Lung Transplant. 2005 Dec;24(12):2262-8. doi: 10.1016/j.healun.2005.07.005. Epub 2005 Nov 17. PMID 16364880
- [Background] Lanuza DM, Lefaiver C, Mc Cabe M, Farcas GA, Garrity E Jr. Prospective study of functional status and quality of life before and after lung transplantation. Chest. 2000 Jul;118(1):115-22. doi: 10.1378/chest.118.1.115. PMID 10893368
- [Background] Linden W, Phillips MJ, Leclerc J. Psychological treatment of cardiac patients: a meta-analysis. Eur Heart J. 2007 Dec;28(24):2972-84. doi: 10.1093/eurheartj/ehm504. Epub 2007 Nov 5. PMID 17984133
- [Background] Mathur S, Reid WD, Levy RD. Exercise limitation in recipients of lung transplants. Phys Ther. 2004 Dec;84(12):1178-87. No abstract available. PMID 15563258
- [Background] Napolitano MA, Babyak MA, Palmer S, Tapson V, Davis RD, Blumenthal JA; Investigational Study of Psychological Intervention in Recipients of Lung Transplant (INSPIRE) Investigators. Effects of a telephone-based psychosocial intervention for patients awaiting lung transplantation. Chest. 2002 Oct;122(4):1176-84. doi: 10.1378/chest.122.4.1176. PMID 12377839
- [Background] Oelberg DA, Systrom DM, Markowitz DH, Zorb SL, Wright C, Wain JC, Ginns LC. Exercise performance in cystic fibrosis before and after bilateral lung transplantation. J Heart Lung Transplant. 1998 Nov;17(11):1104-12. PMID 9855450
- [Background] Tegtbur U, Busse MW, Jung K, Pethig K, Haverich A. Time course of physical reconditioning during exercise rehabilitation late after heart transplantation. J Heart Lung Transplant. 2005 Mar;24(3):270-4. doi: 10.1016/j.healun.2003.12.010. PMID 15737752
- [Background] Van Der Woude BT, Kropmans TJ, Douma KW, Van Der Bij W, Ouwens JP, Koeter GH, Van Der Schans CP. Peripheral muscle force and exercise capacity in lung transplant candidates. Int J Rehabil Res. 2002 Dec;25(4):351-5. doi: 10.1097/00004356-200212000-00014. No abstract available. PMID 12451312
- [Derived] Gutierrez-Arias R, Martinez-Zapata MJ, Gaete-Mahn MC, Osorio D, Bustos L, Melo Tanner J, Hidalgo R, Seron P. Exercise training for adult lung transplant recipients. Cochrane Database Syst Rev. 2021 Jul 20;7(7):CD012307. doi: 10.1002/14651858.CD012307.pub2. PMID 34282853